CLINICAL TRIAL: NCT02585869
Title: A 12-Week, Double-Blind, Placebo-Controlled, Randomized, Multicenter Study to Determine the Efficacy and Safety of CI-1027 in Patients With Low HDL-C and Either Normal or Elevated Triglycerides
Brief Title: Efficacy and Safety of Gemcabene in Patients With Low HDL-C and Either Normal or Elevated Triglycerides
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroBo Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1027-004
Record Dates: First submitted 2015-10-22; First posted 2015-10-23 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Hypercholesterolemia; Hypertriglyceridemia
Keywords: Lipid Regulator; TG
MeSH Terms: conditions — Hypercholesterolemia; Hypertriglyceridemia | interventions — gemcabene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Gemcabene 150 mg (Experimental): Gemcabene 150 mg once daily (QD)
  Interventions: Drug: Gemcabene 150 mg
- Gemcabene 300 mg (Experimental): Gemcabene 300 mg once daily (QD)
  Interventions: Drug: Gemcabene 300 mg
- Gemcabene 600 mg (Experimental): Gemcabene 600 mg once daily (QD)
  Interventions: Drug: Gemcabene 600 mg
- Gemcabene 900 mg (Experimental): Gemcabene 900 mg once daily (QD)
  Interventions: Drug: Gemcabene 900 mg
- Placebo (Placebo Comparator): Placebo once daily (QD)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gemcabene 150 mg — Blinded capsules and tablets, 150 mg, once daily, 84 days
  Arms: Gemcabene 150 mg
Drug: Gemcabene 300 mg — Blinded capsules and tablets, 300 mg, once daily, 84 days
  Arms: Gemcabene 300 mg
Drug: Gemcabene 600 mg — Blinded capsules and tablets, 600 mg, once daily, 84 days
  Arms: Gemcabene 600 mg
Drug: Gemcabene 900 mg — Blinded capsules and tablets, 900 mg, once daily, 84 days
  Arms: Gemcabene 900 mg
Drug: Placebo — Blinded capsule and tablets, once daily, 84 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of gemcabene on HDL-C, LDL-C, TG, and other lipid levels in patients with low HDL-C

ELIGIBILITY:
Inclusion Criteria:

* Men or naturally postmenopausal or surgically menopausal women
* 18 to 80 years of age
* Baseline HDL-C <35 mg/dL (0.9 mmol/L)

Exclusion Criteria:

* Creatine phosphokinase (CPK) >3 × the upper limit of normal (ULN)
* Body Mass Index (BMI) >35 kg/m2
* Uncontrolled Hypertension >95 mm Hg
* Uncontrolled diabetes mellitus (HbA1c >10%)
* Renal dysfunction (blood urea nitrogen [BUN] or creatinine >2 × ULN);
* Hepatic dysfunction (aspartate aminotransferase [AST] or alanine aminotransferase [ALT] >2 × ULN)
* Uncontrolled hypothyroidism (TSH >1.5 × ULN)
* Myocardial infarction, severe or unstable angina pectoris, coronary angioplasty, coronary artery bypass graft, or any other major cardiovascular event resulting in hospitalization in previous 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 1999-12; Primary Completion 2001-06 (Actual); Study Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
HDL-C - percent change from baseline | 84 days

SECONDARY OUTCOMES:
Plasma lipids (eg, LDL-C, VLDL-C, TG)- percent change from baseline | 84 days
Adverse Events | 84 days
Clinical Laboratory - hematology, chemistry, urinalysis | 84 days
  Clinical Laboratory Abnormalities

REFERENCES:
- [Background] Bays HE, McKenney JM, Dujovne CA, Schrott HG, Zema MJ, Nyberg J, MacDougall DE; Gemcabene Study Group. Effectiveness and tolerability of a new lipid-altering agent, gemcabene, in patients with low levels of high-density lipoprotein cholesterol. Am J Cardiol. 2003 Sep 1;92(5):538-43. doi: 10.1016/s0002-9149(03)00721-5. PMID 12943873